CLINICAL TRIAL: NCT02700867
Title: A Randomized Crossover Cadaver Trial Comparing Proximal Tibia and Proximal Humerus Infusion Rates Using the NIO Intraosseous Device During Simulated Cardiopulmonary Resuscitation Performed by Paramedics
Brief Title: Trial Comparing Proximal Tibia and Proximal Humerus Infusion Rates Using the NIO Intraosseous Device
Acronym: IOACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02.006.1MR
Record Dates: First submitted 2016-02-15; First posted 2016-03-07 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Intraosseous Access; Resuscitation
Keywords: intraosseous access; cardiopulmonary resuscitation; paramedic; simulation; cadaver
MeSH Terms: conditions — Cadaver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proximal tibia (Experimental): Assumption of intraosseous access into the proximal tibia. Simulation of continous resuscitation was carried out using a system of chest compression LifeLine ARM.
  Interventions: Device: NIO
- Proximal humerus (Experimental): Assumption of intraosseous access into the proximal humerus. Simulation of continous resuscitation was carried out using a system of chest compression LifeLine ARM.
  Interventions: Device: NIO

INTERVENTIONS:
Device: NIO — Intraosseous access device NIO (Defibtech)

SUMMARY:
The investigators sought to compare the intraosseous access success rates of the proximal tibia and the proximal humerus using new Intraosseous access device "NIO" in an adult cadaver model during simulated resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* paramedics
* without previous experience in intraosseous devices

Exclusion Criteria:

* not meet the above criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Success rate | 1 day
  Success rate of IO cannulation was defined as successful administration of infusion solutions via the performed IO access. Failure was defined as extravasation or unsuccessful (first) effort of IO insertion.

SECONDARY OUTCOMES:
Time of IO insertion | 1 day
  Procedure time was defined as the duration of picking up the prepared set of IO device from the shelf, preparation of the access set and patients' insertion site including disinfection and draping, insertion procedure of the cannula itself, assembling of the access set and first successful administration of drugs or infusion solutions through the newly established vascular access. The time taken for each infusion attempt was measured offline while reviewing procedures by videotape, and subsequently entered into a computer spreadsheet. Times were measured in seconds.
Ease-of-use | 1 day
  ease-of-use of the NIO in tibia and humerus using a five-point Likert Scale ("the device is easy to use"; 1-strongly disagree, 2-disagree, 3-neither agree nor disagree, 4-agree, 5-strongly agree).
first location | 1 day
  Participants were asked to record their "first location access" tibia or humerus

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szarpak L, Truszewski Z, Smereka J, Krajewski P, Fudalej M, Adamczyk P, Czyzewski L. A Randomized Cadaver Study Comparing First-Attempt Success Between Tibial and Humeral Intraosseous Insertions Using NIO Device by Paramedics: A Preliminary Investigation. Medicine (Baltimore). 2016 May;95(20):e3724. doi: 10.1097/MD.0000000000003724. PMID 27196493